CLINICAL TRIAL: NCT01569399
Title: Evaluation de l'efficacité thérapeutique de la Stimulation magnétique transcrânienne répétée Sur le Traitement du Craving à l'Alcool et la prévention de la Rechute Alcoolique à 6 Mois Chez Les Sujets dépendants et Des Facteurs génétiques déterminant la réponse thérapeutique
Brief Title: Efficacity of rTMS in Alcohol Dependance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10-21; 2010-A00727-32 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-03-14; First posted 2012-04-03 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Alcohol Dependance
Keywords: Alcohol dependance; rTMS; craving; alcohol consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active rTMS (Active Comparator): High frequency (10HZ) on the left DLPFC
  Interventions: Other: rTMS (repetitive transcranial magnetic stimulation)
- sham rTMS (Placebo Comparator)
  Interventions: Other: rTMS (repetitive transcranial magnetic stimulation)

INTERVENTIONS:
Other: rTMS (repetitive transcranial magnetic stimulation) — Frequency (10hz) 120% motor threshold 10 sessions

SUMMARY:
Prior research in substance dependence has suggested potential anti-craving effects of repetitive transcranial magnetic stimulation (rTMS) when applied to the dorsolateral prefrontal cortex (DLPFC). The aim of the investigators study was to investigate the effect of high frequency rTMS of the left dorsolateral prefrontal cortex compared to sham stimulation on craving and alcohol consumption.

DETAILED DESCRIPTION:
Prior research in substance dependence has suggested potential anti-craving effects of repetitive transcranial magnetic stimulation (rTMS) when applied to the dorsolateral prefrontal cortex (DLPFC). The aim of our study was to investigate the effect of high frequency rTMS of the left dorsolateral prefrontal cortex compared to sham stimulation on craving and alcohol consumption.

150 detoxified patients are randomized either to a high frequency rTMS over the left DLPFC (n = 75) or a sham stimulations (n = 75). Alcohol craving is determined with the Obsessive Compulsive Drinking Scale. Patients are allocated to active and sham rTMS in a 1: 1 ratio, such that 75 patients received active and 75 patients sham rTMS to the left DLPFC (10 Hz frequency, total 10 sessions). The Alcohol Craving Questionnaire (ACQ-NOW) and the Obsessive Compulsive Drinking Scale (OCDS) are administered to measure the severity of alcohol craving at baseline, after the last rTMS session and day 15, M1, M3, M6 after. Alcohol drinking is evaluated with Timeline Followback (TLFB).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcohol dependence syndrome according to DSM-IV criteria
* Detoxified inpatients hospitalised for Alcohol Withdrawal for more than one week
* Giving written informed

Exclusion Criteria:

* Left-handed patients at the time of inclusion.
* Age < 18 years
* Withdrawal Assessment (CIWA-Ar) scores of > 5
* Patients with major medical or neurological disorders or with a pacemaker or metal in any part of the body were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Superiority of left rTMS (DLPFC)on reduction of alcohol consumption in AD patients compared to sham rTMS | Patients will be followed during 6 month
  Evaluation of the intensity of craving (AUQ, Borg analogic scale, OCDS) and total day with no alcohol use measured with TLFB at Day 0, Day 5, Day 15, Month1 , Month3 and Month6 in AD outpatients.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DUBERTRET, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Louis Mourier Hospital, Colombes, France